CLINICAL TRIAL: NCT05957510
Title: Evaluation of Safety and Efficacy of Serplulimab Plus Chemotherapy in Patients With Histological Transformation From EGFR-mutated NSCLC to SCLC After Treatment: a Single-arm, Multicenter, Open-label Phase II Study
Brief Title: Safety and Efficacy Evaluation of Serplulimab Plus Chemo in SCLC Transformed From EGFR-mutated NSCLC After Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jin-Ji Yang, Principal Investigator, Guangdong Association of Clinical Trials
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2302 (HLX10IIT39)
Record Dates: First submitted 2023-07-05; First posted 2023-07-24 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Small-cell Lung Cancer
Keywords: transformed SCLC, EGFR-mutated NSCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Patients who met the inclusion criteria, did not meet the exclusion criteria, and agreed to accept the treatment plan of this study will undertake a combination chemotherapy regimen, comprised of serplulimab (300mg), etoposide (100 mg/m2), and carboplatin (AUC 5 mg/mL/min, up to 750mg). These agents will be administered intravenously in 3-week intervals over a span of 4 to 6 cycles.
  Interventions: Drug: Serplulimab
- Cohort 2 (Experimental): Patients who met the specific inclusion criteria, did not meet the specific exclusion criteria, and agreed to accept the treatment of this study will undertake the same treatment as cohort 1 in the form of ' compassionate use '.
  Interventions: Drug: Serplulimab
- Cohort 3 (Experimental): Patients with treatment contraindications or unwillingness to accept the treatment of this study will be treated with the clinical routine treatment recommended by the investigator.
  Interventions: Drug: SOC

INTERVENTIONS:
Drug: Serplulimab — serplulimab 300mg, d1, q3w, iv. etoposide 100 mg/m2, d1-3, q3w, iv. carboplatin AUC 5 (up to 750mg), d1, q3w, iv.
  Other Names: etoposide; carboplatin
  Arms: Cohort 1; Cohort 2
Drug: SOC — the treatment recommended by the investigator
  Arms: Cohort 3

SUMMARY:
This investigator-initiated, open-label, prospective Phase II clinical trial, planned to take place across multiple centers in China. We design this trial to evaluate the safety and efficacy of Serplulimab plus chemotherapy in SCLC transformed from EGFR-mutated NSCLC after treatment.

DETAILED DESCRIPTION:
Participants with EGFR-mutant NSCLC who were transformed into SCLC after treatment and did not undergo systemic anticancer therapy after transformation will be divided into three cohorts. We plan to enroll 36 patients in the first cohort, and 18 patients in the second cohort. Participants in cohort 1 and cohort 2 will undertake a combination chemotherapy regimen, comprised of serplulimab (300mg), etoposide (100 mg/m2), and carboplatin (AUC 5 mg/mL/min, up to 750mg). These agents will be administered intravenously in 3-week intervals over a span of 4 to 6 cycles. Participants in cohort 3 will be treated with the clinical routine treatment recommended by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in clinical studies.
* Age 18-75 (including the cut-off value) when signing the Informed Consent Form (ICF)
* Patients must provide pathological diagnosis reports and genetic testing reports before transformation, and the reports clearly indicate that they were non-small cell lung cancer containing EGFR mutations before transformation.
* Patients must provide a pathological diagnosis report after transformation, as well as 10 unstained reports after transformation. The pathology of the patients after transformation was SCLC or high-grade neuroendocrine carcinoma or containing SCLC components.
* Patients who have not received systemic therapy and anti-PD-1/L1 and CTLA-4 therapy after tissue type transformation. Patients are allowed to receive immunotherapy before transformation, but the last line of therapy cannot contain immunotherapy.
* The end of previous anti-tumor treatment must be more than 2 weeks from the first medication in this study, and the treatment-related AE should be recovered to CTCAE 5.0 ≤ grade 1 (except for grade 2 alopecia).
* At least one measurable target lesion based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria identified within the four weeks leading up to the initial treatment dose
* ECOG PS 0 or 1
* Expected life expectancy of 12 weeks or more
* Adequate organ function
* The serum pregnancy test of female patients must be negative within 14 days before treatment, and effective contraceptive measures should be taken during treatment and within 6 months after treatment. Lactation is prohibited during treatment.
* Male patients must agree to abstinence (avoid heterosexual intercourse) or take contraceptive measures.

Exclusion Criteria:

* Patients cannot provide a pathology report after tissue type transformation.
* Patients with a known history of severe allergies to any monoclonal antibody ( NCI-CTCAE 5.0 grade greater than grade 3 ); or known hypersensitivity to carboplatin/etoposide components.
* Patients with known or screening findings of active central nervous system (CNS) metastases and/or cancerous meningitis (Exceptions will be made for patients with asymptomatic brain metastases or those who have had stable brain metastases for at least 4 weeks after treatment)
* Patients who have received systemic therapy or other immune checkpoint inhibitors after tissue type transformation; patients who are preparing for or have previously received organ or bone marrow transplantation.
* Any active infection requiring systemic anti-infectious therapy within 14 days before the first administration.
* Myocardial infarction or poorly controlled arrhythmia has occurred within 6 months before the first administration; or according to the NYHA standard III-IV cardiac insufficiency or echocardiography left ventricular ejection fraction < 50 %; or pleural effusion, pericardial effusion or ascites requiring clinical intervention.
* Patients have uncontrolled or symptomatic hypercalcemia; Patients have poor blood pressure control; patients with deep vein thrombosis, being treated with anticoagulant or platelet therapy, or previous deep vein thrombosis or severe bleeding caused by the use of anti-angiogenic drugs; Patients with known active or suspected autoimmune diseases (Patients in a stable state who do not require systemic immunosuppressive therapy are allowed to be enrolled).
* Patients who have been and were screened and judged by the investigator to be likely to interfere with the detection and management of suspected drug-related lung toxicity; Patients who the investigator believes have any factors that are inappropriate for participating in this trial.
* Patients with hepatitis B; or hepatitis C patients; or syphilis screening positive; or known human immunodeficiency virus ( HIV ) positive history or HIV screening positive; known history of mental drug abuse or drug abuse.
* Other active malignancies tumors within 5 years or concurrently.
* Patients who were vaccinated with live or attenuated vaccines within 28 days before the first dose, or had plans to vaccinate such vaccines during the study period (but inactivated virus vaccines for seasonal influenza are allowed) or who underwent major surgery.
* Patients with spinal cord compression who have not been radically cured by surgery and/or radiotherapy. Received radical radiotherapy within 3 months before the first administration.
* Patients who were participating in other clinical studies, or who participated in any other clinical trials (including drugs and devices, etc.) and received intervention within 3 months or 5 half-lives (whichever is longer) before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From date of first dosing to first documented progression or death from any cause, whichever came first, assessed up to 2 years.
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST v1.1).

SECONDARY OUTCOMES:
Objective Response Rate | Up to 2 years
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.
Overall survival (OS) | Up to approximately 2 years
  OS is the time from the date of first dosing date to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ji Yang, PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial Perople's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang J, Zhang XH, Cai Y, Yang D, Shi J, Xing P, Xu T, Wu L, Su W, Xu R, Wei T, Chen HJ, Yang JJ. Rationale and Design of a Phase II Trial of Combined Serplulimab and Chemotherapy in Patients with Histologically Transformed Small Cell Lung Cancer: a Prospective, Single-arm and Multicentre Study. Clin Oncol (R Coll Radiol). 2024 Jan;36(1):39-45. doi: 10.1016/j.clon.2023.11.030. Epub 2023 Nov 11. PMID 37977903